CLINICAL TRIAL: NCT03878095
Title: A Phase II Study of Olaparib and AZD6738 in Isocitrate Dehydrogenase (IDH) Mutant Solid Tumors
Brief Title: Testing Olaparib and AZD6738 in IDH1 and IDH2 Mutant Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-01461; NCI-2019-01461 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2000027026; 10222 (Other: Yale University Cancer Center LAO); 10222 (Other: CTEP); UM1CA186689 (NIH)
Record Dates: First submitted 2019-03-15; First posted 2019-03-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Malignant Solid Neoplasm; Refractory Cholangiocarcinoma; Refractory Malignant Solid Neoplasm
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Biopsy; Specimen Handling; ceralasertib; Magnetic Resonance Spectroscopy; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (olaparib, ceralasertib) (Experimental): Patients receive olaparib PO BID on days 1-28 of each cycle and ceralasertib PO QD on days 1-7 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsies during screening and on study, collection of blood samples throughout the trial, and undergo CT and/or MRI scans throughout the trial. Patients may also undergo bone marrow aspiration and biopsy as clinically indicated on study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Bone Marrow Aspiration; Procedure: Bone Marrow Biopsy; Drug: Ceralasertib; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging; Drug: Olaparib

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsies
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspiration and biopsy
Procedure: Bone Marrow Biopsy — Undergo bone marrow aspiration and biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Drug: Ceralasertib — Given PO
  Other Names: AZD6738
Procedure: Computed Tomography — Undergo CT scans
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI scans
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU 0059436; KU-0059436; KU0059436; Lynparza; Olanib; Olaparix; PARP Inhibitor AZD2281

SUMMARY:
This phase II trial studies how well olaparib and ceralasertib (AZD6738) work in treating patients with IDH mutant cholangiocarcinoma or solid tumors. Cancer is caused by changes (mutations) to genes that control the way cells function. Laboratory studies have shown that olaparib and AZD6738 can shrink IDH mutant tumors or stop them from growing. Olaparib and ceralasertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the overall response rates of olaparib and ceralasertib (AZD6738) in subjects with recurrent/progressive IDH1/2-mutant solid malignant tumors, who will be recruited to 2 cohorts:

Ia. Cholangiocarcinoma (cohort has been closed to accrual); Ib. Other solid malignant tumors.

SECONDARY OBJECTIVES:

I. To assess the progression free survival (PFS) of olaparib and AZD6738 in adults with recurrent/progressive IDH1/2-mutant solid malignant tumors.

II. To estimate the overall survival (OS) in adults with recurrent/progressive IDH1/2- mutant solid malignant tumors.

III. To assess the duration of response in adults with recurrent/progressive IDH1/2-mutant solid malignant tumors.

IV. To assess the safety and tolerability of the combination of olaparib and AZD6738.

EXPLORATORY OBJECTIVES:

I. To evaluate 2-hydroxyglutarate (2HG) concentration in plasma by mass spectrometry and correlate with treatment response.

II. To evaluate 2HG levels in tumor biopsies prior to the beginning of treatment and while on therapy and correlate with treatment response.

III. Correlate 2HG concentration in plasma and in tumor biopsies. IV. To evaluate deoxyribonucleic acid (DNA) double strand breaks (DSBs) as measured by mass cytometry time of flight (CyTOF)-imaging mass cytometry (IMC) in tumor biopsies before and after treatment with olaparib and AZD6738.

OUTLINE:

Patients receive olaparib orally (PO) twice daily (BID) on days 1-28 of each cycle and ceralasertib PO once daily (QD) on days 1-7 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsies during screening and on study, collection of blood samples throughout the trial, and undergo computed tomography (CT) and/or magnetic resonance imaging (MRI) scans throughout the trial. Patients may also undergo bone marrow aspiration and biopsy as clinically indicated on study.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand the nature of this trial and provide written informed consent, prior to any study specific procedures. Patients with impaired decision making capacity (IDMC) who have a close caregiver or legally authorized representative (LAR) may be considered eligible for this study at the treating physician's discretion, provided that the physician is reasonably sure that the possible risks and benefits of the study are clear and that the patient will take the drug as prescribed
* Subjects must be diagnosed with a solid malignant tumor (other than cholangiocarcinoma or primary central nervous system [CNS] tumor) that has progressed despite standard therapy, or for which no effective standard therapy exists. Patients with cholangiocarcinoma are no longer allowed as this cohort has closed to accrual. Patients with primary CNS tumors, e.g. glioma, are not allowed
* Patients must have biopsy-confirmed evidence of an IDH1 or IDH2 mutation, confirmed in a Clinical Laboratory Improvement Act (CLIA)-certified laboratory, associated with neomorphic activity of the encoded proteins
* Patients must have tumors determined to be easily accessible for biopsy and must be willing to have serial biopsies. Tumor biopsies will be performed on the most accessible biopsiable site of disease. All possible precautions to avoid complications will be taken, including discussions in multidisciplinary meetings, if needed. If a patient opts out of a pre-treatment biopsy, biopsy is not possible, or if a pre-treatment biopsy does not yield sufficient tissue for analysis, the patient must be willing to provide a sufficient archival formalin-fixed paraffin-embedded (FFPE) specimen for liquid chromatography/mass spectrometry (LC/MS) analysis of 2HG in order to enroll on the study. Permission of the study principal investigator (PI) is required in all of the above scenarios

  * In order to maximize the availability of newly obtained specimens for 2-HG analysis, at least 10 biopsies will be required in each group (cholangiocarcinoma and other solid tumors) of 14 patients treated in the first stage of this Simon two-stage design. Thus if 4 patients in an arm have already opted out, further patients may only enroll on that arm (in the first stage) if they agree to undergo the pre- and on-treatment biopsies. If a patient has agreed to undergo the two biopsies and undergoes the pre-treatment biopsy, he or she may not opt out of the second biopsy unless such a biopsy would not be safe (e.g. inaccessible tumor). Permission of the study PI is required in this scenario
  * All patients must be willing to provide 5 unstained archival slides, if available, for pre-treatment 2-HG analysis and correlation with 2-HG levels in pre-treatment frozen specimens
* Patients must be willing to undergo extra blood sampling for correlative studies
* Patients must have measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
* Patients must have at least one lesion, not previously irradiated, that can be accurately measured at baseline as >= 10 mm in the longest diameter (except lymph nodes which must have short axis >= 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) or >= 10 mm with callipers by clinical exam OR at least one lesion (measurable) that can be accurately assessed by CT/MRI/clinical exam at baseline and follow up visits
* Subjects must have progressive cancer at the time of study entry
* Prior experimental (non-Food and Drug Administration [FDA] approved) therapies (other than drugs that target ATR) and immunotherapies are allowed. Patients must not have received these therapies for 30 days or five half-lives of the drug (whichever is less) prior to the initiation of study treatment
* Toxicities from prior therapies should have recovered to =< grade 1, with the exception of stable chronic grade 2 toxicities that are not overlapping with presumed toxicities of olaparib
* Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after central nervous system (CNS)-directed treatment, as ascertained by clinical examination and brain imaging (MRI or CT scan) during the screening period
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required for at least 4 weeks (or scheduled assessment after the first cycle of treatment), and a risk-benefit analysis (discussion) by the patient and the investigator favors participation in the clinical trial
* If evidence of chronic hepatitis B virus (HBV) infection, HBV viral load must be undetectable on suppressive therapy if indicated. If history of hepatitis C virus (HCV) infection, must be treated with undetectable HCV viral load
* Female/male of age >= 18 years. This is because no dosing or adverse event data are currently available on the use of olaparib or AZD6738 in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG) 0-1 (Karnofsky >= 70%)
* Hemoglobin >= 10.0 g/dL with no blood transfusion in < 14 days prior to starting therapy (measured within 14 days prior to administration of study treatment)
* Leukocytes >= 3,000/mcL (measured within 14 days prior to administration of study treatment)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (measured within 14 days prior to administration of study treatment)
* Platelet count >= 100 x 10^9/L (measured within 14 days prior to administration of study treatment)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (measured within 14 days prior to administration of study treatment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamic pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal unless liver metastases are present in which case they must be =< 5 x ULN (measured within 14 days prior to administration of study treatment)
* Creatinine clearance estimated using the Cockcroft-Gault equation of >= 51 mL/min or based on a 24 hour urine test (measured within 14 days prior to administration of study treatment)
* No features suggestive of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML) on peripheral blood smear when performed as clinically indicated
* Patients must have a life expectancy of >= 16 weeks, in the opinion of the treating physician
* Patients must be willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Prior radiation therapy is allowed. Patients must not have received radiation therapy within 3 weeks prior to the initiation of study treatment
* Women of child-bearing potential are expected to use highly effective contraception during the study and for 6 months after the last dose of study drug. Postmenopausal or evidence of non-childbearing status for women of childbearing potential: negative urine or serum pregnancy test within 28 days of study treatment and confirmed prior to treatment on day 1

  * Postmenopausal is defined as:

    * Amenorrheic for 1 year or more following cessation of exogenous hormonal treatments
    * Luteinizing hormone (LH) and follicle stimulating hormone (FSH) levels in the post-menopausal range for women under 50
    * Radiation-induced oophorectomy with last menses > 1 year ago
    * Chemotherapy-induced menopause with > 1 year interval since last menses
    * Surgical sterilization (bilateral oophorectomy or hysterectomy)
* Male patients and their partners, who are sexually active and of childbearing potential, must agree to the use of two highly effective forms of contraception in combination, throughout the period of taking study treatment and for 6 months after last dose of study drug(s) to prevent pregnancy in a partner
* Patients with human immunodeficiency virus (HIV) on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study
* Previous enrollment in the present study
* Participation in another clinical study with an investigational product during the last 30 days or five half-lives of the drug (whichever is less) prior to the initiation of study treatment
* Any previous treatment with a PARP inhibitor
* Any previous treatment with AZD6738 or any other ATR inhibitor
* Patients receiving any systemic chemotherapy or radiotherapy within 3 weeks prior to study treatment
* Other malignancy within the last 5 years except: adequately treated non-melanoma skin cancer, curatively treated in situ cancer of the cervix, ductal carcinoma in situ (DCIS), stage 1, grade 1 endometrial carcinoma, or other solid tumors including lymphomas (without bone marrow involvement) curatively treated with no evidence of disease for >= 5 years. Patients with a history of localized triple negative breast cancer may be eligible, provided they completed their adjuvant chemotherapy more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Resting electrocardiography (ECG) indicating uncontrolled, potentially reversible cardiac conditions, as judged by the investigator (e.g., unstable ischemia, uncontrolled symptomatic arrhythmia, congestive heart failure, Fridericia's corrected QT [QTcF] prolongation > 500 ms, electrolyte disturbances, etc.), or patients with congenital long QT syndrome
* Concomitant use of known strong CYP3A inhibitors (e.g. itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir) or moderate CYP3A inhibitors (e.g. ciprofloxacin, erythromycin, diltiazem, fluconazole, verapamil). The required washout period prior to starting study treatment is 2 weeks
* Concomitant use of known strong (e.g. phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) or moderate CYP3A inducers (e.g. bosentan, efavirenz, modafinil). The required washout period prior to starting study treatment is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents
* Persistent toxicities caused by previous cancer therapy. Toxicities should have recovered to =< grade 1, excluding alopecia, or should be stable chronic grade 2 toxicities that do not overlap with presumed toxicities of olaparib and/or AZD6738
* Patients with myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML) or features suggestive of MDS/AML
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are not eligible if the treating physician determines that immediate CNS specific treatment is required, and a risk-benefit analysis (discussion) by the patient and the investigator does not favor participation in the clinical trial. A scan to confirm the absence of brain metastases is not required. The patient can receive a stable dose of corticosteroids before and during the study if these were started at least 4 weeks prior to treatment. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 28 days
* Major surgery within 2 weeks of starting study treatment. Major surgeries typically require general anesthesia, are associated with an estimated blood loss of > 500 mL, and require an overnight hospital stay. Examples include laparoscopic surgery, open resection of organs, joint replacements and other orthopedic surgeries, and vascular or intracranial surgeries. Examples of minor surgeries include those performed on an ambulatory basis, cataract surgery, dental surgeries, cutaneous, endoscopic, and arthroscopic procedures. Effects from major surgeries should have recovered to =< grade 1, with the exception of stable chronic grade 2 toxicities that are not overlapping with presumed toxicities of olaparib and/or AZD6738
* Patients considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 3 months) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, extensive interstitial bilateral lung disease on high resolution computed tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent and would limit compliance with study requirements
* Patients unable to swallow orally administered medication and patients with gastrointestinal disorders likely to interfere with absorption of the study medication
* Women who are actively breast feeding
* Patients with a known hypersensitivity to olaparib or AZD6738 or any of the excipients of the products. History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib or AZD6738
* Previous allogeneic bone marrow transplant or double umbilical cord blood transplantation (dUCBT)
* Whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable within the last 28 days)
* Patients who are receiving any other investigational agents
* Pregnant women are excluded from this study because olaparib is an agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with olaparib, breastfeeding should be discontinued if the mother is treated with olaparib
* Receiving, or having received during the 14 days prior to first dose, corticosteroids (at a dose > 10 mg prednisone/day or equivalent) for any reason
* Any of the following cardiac diseases currently or within the last 6 months (by New York Heart Association [NYHA] >= class 2 where applicable):

  * Unstable angina pectoris
  * Congestive heart failure or known reduced left ventricular ejection fraction (LVEF) < 55%
  * Acute myocardial infarction
  * Conduction abnormality not controlled with pacemaker or medication e.g. complete left bundle branch block, third degree heart block
  * Significant ventricular or supraventricular arrhythmias e.g. (patients with chronic rate-controlled atrial fibrillation in the absence of other cardiac abnormalities are eligible)
* Patients at risk of brain perfusion problems, e.g., medical history of carotid stenosis or pre-syncopal or syncopal episodes, history of transient ischemic attacks (TIAs)
* Uncontrolled hypertension (grade 2 or above) requiring clinical intervention
* Any factors that increase the risk of corrected QT (QTc) prolongation or risk of arrhythmic events such as congestive heart failure, unstable angina pectoris, acute myocardial infarction, hypokalemia, congenital long QT syndrome, immediate family history of long QT syndrome or unexplained sudden death under 40 years of age, conduction abnormality not controlled with pacemaker or medication
* Patients with relative hypotension (< 90/60 mm Hg) or clinically relevant orthostatic hypotension, including a fall in blood pressure of > 20 mm Hg
* Refractory nausea and vomiting, chronic gastrointestinal diseases or previous significant bowel resection, with clinically significant sequelae that would preclude adequate absorption of AZD6738

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-30 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 30 days post treatment after removal from study
  The exact two-sided 95% confidence intervals (CIs) for the ORR will be reported.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From start of treatment to time of progression or death, whichever occurs first, assessed up to 30 days after removal from study
  PFS will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on the Greenwoods variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease on the survival data. The adjusted p-values of the odds ratios and the adjusted 95% confidence interval will be reported.
Overall survival (OS) | From start of treatment to time of death, assessed up to 30 days after removal from study
  OS will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on the Greenwoods variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease on the survival data. The adjusted p-values of the odds ratios and the adjusted 95% confidence interval will be reported.
Duration of response | From the time measurement criteria are met for complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 30 days after removal from study
  Will be estimated using the Kaplan-Meier method with the 95% CIs. The CI based on the Greenwoods variance will be reported. In addition, the possible risk factors will be compared for survival with log-rank test. For multivariate analysis, the proportional hazards Cox model will be applied to investigate potential prognostic factors, such as age and stage of disease on the survival data. The adjusted p-values of the odds ratios and the adjusted 95% confidence interval will be reported.
Incidence of adverse events | Up to 30 days post treatment
  Toxicities will be evaluated utilizing the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0.

OTHER OUTCOMES:
Absolute and fold changes in gamma H2AX foci | Baseline up to 30 days post treatment
  Absolute and fold changes for gamma H2AX foci will be calculated between baseline and subsequent follow-up (pre-treatment and on-treatment biopsies). These will be displayed graphically versus (vs.) time for each cohort. Differences will be plotted vs. response status. Wilcoxon sign-rank test as well as paired t-tests will be used to evaluate if differences between baseline and each subsequent time point are significant. Summary statistics will be reported (with 95% confidence intervals) to demonstrate mean differences in fold-change (or log fold-change) between responders and non-responders.
2HG levels | Up to 30 days post treatment
  2HG levels in tumor and plasma will be compared to treatment responses. The Mann-Whitney U test will be used to test for differences in post-treatment tissue and plasma 2HG concentrations between patients with a response to treatment and those without. Will also apply analysis of covariance for post-treatment plasma concentration in 2HG adjusted for the pre-treatment plasma concentration between patients with a response to treatment and those without.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M LoRusso, Principal Investigator — Yale University Cancer Center LAO
Locations (13):
- United States (13):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-08-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03878095/ICF_000.pdf